CLINICAL TRIAL: NCT01463592
Title: An Open Labelled, Active Controlled, Three Arm, Parallel- Group Study of the Safety and Efficacy of Renessans Administered Alone and in Combination With Standard Interferon Therapy in Patients Chronic HCV Hepatitis
Brief Title: To Study the Efficacy and Safety of Renessans in Chronic HCV Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MTI Medical Private Limited, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REN1
Record Dates: First submitted 2011-08-30; First posted 2011-11-02 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-10

CONDITIONS: Hepatitis C, Chronic
Keywords: Renessans; HCV
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Interferon alpha-2; Ribavirin; viron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group II a (Experimental): TRIPPLE THERAPY
  Interventions: Biological: RENESSANS , INTERFERON ALPHA 2b, Ribavirin
- Group II b (Active Comparator): DUAL THERAPY
  Interventions: Drug: Interferon Alfa-2b AND RIBAVIRIN
- Group I (Experimental): ORAL RENESSANS
  Interventions: Biological: RENESSANS

INTERVENTIONS:
Biological: RENESSANS , INTERFERON ALPHA 2b, Ribavirin — ORAL RENESSANS 5gm. Twice Daily +INTERFERON ALPHA 2b 3 Million Units s/c +RIBAVIRIN 15mg/kg
  Other Names: IODINE POLYMER; HEBERON; VIRON
  Arms: Group II a
Drug: Interferon Alfa-2b AND RIBAVIRIN — INTERFERON ALPHA 2b 3 Million Units s/c +RIBAVIRIN 15mg/kg
  Other Names: HEBERON; VIRON
  Arms: Group II b
Biological: RENESSANS — ORAL RENESSANS 5gm. Thrice Daily{active iodine 300mg} for 6months
  Other Names: IODINE POLYMER
  Arms: Group I

SUMMARY:
Chronic HCV infection is one of the common causes of the chronic liver disease. Approximately 6-10% of the general public is expected to be suffering from this infection. In case that these patients are not treated at an appropriate time, these patients develop the sequelae of the chronic liver disease e.g. cirrhosis of liver, Ascites, and Hepatocellular carinoma. Interferon alpha 2 a or alpha 2b injections and Ribavirin combination is the treatment of choice for people suffering from Chronic HCV infection and this combination need to be administered for 6-12 months. Interferons are biological agents and are to be administered parenterally. Interferons are expensive and are associated with number of minor and major adverse effects. Ribavirin is also associated with significant adverse effects. These compounds cannot be considered as one of the ideal forms of the treatment.

In the past, quite a few natural products have been tested to assess their hepatoprotective activity and possibly anti viral activity as well. These include Vitamin C (Ascorbic acid), Vitamin E, Zinc, Silymarin, Red beet roots, crushed licorice and etc. etc.

Rationale Iodine , Potassium iodide and Ascorbic acid are natural products used in the management of Thyroiditis and chronic cutaneous fungal infections. This combination of iodine compounds along with ascorbic acid is being used for the management of chronic hepatitis B & C in the central Asian states e.g. Kazakhstan etc.

The investigators have conducted a feasibility study in which oral Iodine Compound {RENESSANS} was given to patients suffering HCV related Chronic Active Hepatitis and anti-viral activity and safety has been analyzed. In this study, RENESSANS containing regimen has been well tolerated by all the patients and has shown some antiviral activity.

In this study the investigators will assess whether the administration of RENESSANS {oral } improves the antiviral activity in patients receiving standard interferon therapy.

DETAILED DESCRIPTION:
1. Primary

   The primary objective of this study is to assess the efficacy of combination therapy comprising of RENESSANS, INTERFERONS and RIBAVIRIN in the management of treatment naïve HCV related Chronic Active Hepatitis patients.
2. Secondary

   The secondary objectives of this study are:
   1. Determine the biochemical or virological improvement in patients suffering from HCV related Chronic Active Hepatitis.
   2. Determine the safety and tolerability of Renessans {oral} when administered as a part of antiviral activity outlined in this protocol.
3. ENDPOINTS

   The primary endpoint will be the number of subjects achieving
   1. Virological response as evident by Rapid Viral Response(RVR), Early Viral Response(EVR) and Sustained Viral Response(SVR).
   2. Biochemical response as evident by normalization of ALT.

   The secondary endpoint will be

   a. Assessment of the safety and tolerability of RENESSANS through: routine physical examination, routine clinical laboratory tests, clinical monitoring and adverse events reporting.
4. INVESTIGATIONAL PLAN

   Study Design.

   This is an open labeled, active controlled, three arm, parallel-group study of the safety and efficacy of the oral formulation of natural iodine compound (Renessans) administered alone and in combination with standard interferon therapy in patient suffering from chronic HCV hepatitis.

   The enrolled patients will be tested for following base line laboratory tests

   VISIT 1:

   CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes Thyroid Function tests HBsAg, HIV antibody Urinalysis ANA, RA factor and serum ferritin levels USG of abdomen HCV RNA (PCR by amplicor, roche) qualitative analysis, if positive then quantitative analysis (Real time) and genotype as well.

   Pregnancy test in case of females Informed consent shall be obtained and each individual patient's treatment risk shall be covered under a certified health insurance plan.

   Renessans will be administered in eligible patients as follows:

   Study Arm Dosing Schema Group I ORAL RENESSANS 5gm. Thrice Daily{active iodine 300mg} for 6months Group II a ORAL RENESSANS 5gm. Twice Daily +INTERFERON ALPHA 2b 3 Million Units s/c +RIBAVIRIN 15mg/kg Group II b INTERFERON ALPHA 2b 3 Million Units s/c +RIBAVIRIN 15mg/kg Blood samples shall be collected and stored for post - hoc analysis of HCV RNA at day 1, 7 and 15(visit 2,3 & 4).

   Patients will be reviewed for the hepatoprotection, anti viral activity and any adverse event every four weeks with following clinical and lab work.

   VISIT 5 Detailed history and physical examination Following lab. Investigations at week 4. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes Thyroid Function tests Ferritin HCV RNA (PCR) quantitative analysis VISIT 6 Detailed history and physical examination Following lab. Investigations at week 8. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes

   VISIT 7 Detailed history and physical examination Following lab. Investigations at week 12. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes Thyroid Function tests Ferritin HCV RNA (PCR) quantitative analysis

   VISIT 8 Detailed history and physical examination Following lab. Investigations at week 16. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes VISIT 9 Detailed history and physical examination Following lab. Investigations at week 20. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes VISIT 10 Detailed history and physical examination Following lab. Investigations at week 24. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes VISIT 11 Detailed history and physical examination Following lab. Investigations at week 28. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes VISIT 12 Detailed history and physical examination Following lab. Investigations at week 32. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes VISIT 13 Detailed history and physical examination Following lab. Investigations at week 36. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes VISIT 14 Detailed history and physical examination Following lab. Investigations at week 40. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes VISIT 15 Detailed history and physical examination Following lab. Investigations at week 44. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes VISIT 16 Detailed history and physical examination Following lab. Investigations at week 48. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes VISIT 15 Detailed history and physical examination Following lab. Investigations at week 52. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes VISIT 15 Detailed history and physical examination Following lab. Investigations at week 60. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes

   VISIT 16 Detailed history and physical examination Following lab. Investigations at week 72. CBC including platelet count and ESR Liver function tests including albumin and total proteins. Creatinine Serum electrolytes Thyroid Function tests Ferritin HCV RNA (PCR) quantitative analysis

ELIGIBILITY:
Inclusion Criteria:

* Following groups of the people will be enrolled for the study.

  * Patients suffering from chronic HCV infection as evident with a positive serology for Anti HCV antibody and raised ALT.
  * Both males and females
  * Age group: 18 - 55 years
  * Informed consent

Exclusion Criteria:

* Following groups of people will be excluded from the study

  * Pregnant females
  * Body mass index more than 25
  * Uncontrolled Diabetes Mellitus, Hypertension, Ischemic heart disease, Renal failure, Respiratory failure, Chronic infections, gall stone disease or renal stone disease.
  * Patients known to have hypersensitivity to Iodine compounds in the past.
  * Psychiatric disorders except mild anxiety disorders.
  * Patients suffering from auto immune diseases e.g. Rheumatoid Arthritis, SLE, or thyroid diseases.
  * Patients suffering from concomitant HBV infection, HIV infection or any other chronic liver disease.
  * Bilirubin more than 2mg/dl, Albumin less than 3.0 gms/dl, INR more than 1.5, Hb. less than 10 gms /dl, absolute neutrophil count less than 1500/cmm and platelet count less than 100,000/cmm
  * Serum sodium less than 130mmol/l.
  * Patients who have received the interferon treatment in the past.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Renessans based triple therapy versus dual therapy | 03 years
  Efficacy will be assessed by biochemical and virological response. Biochemical response will be assessed in the form of mean decline in ALT from baseline at 3 month and end of treatment. Virological response will be assessed in the form of response guided therapy i-e RVR [negative RNA at week 4],EVR [negative RNA at 12 weeks],ETR [negative RNA at end of treatment] and SVR[negative PCR after 6 month of completion of therapy].

SECONDARY OUTCOMES:
Assess the safety and tolerability of Renessans in patients with chronic HCV patients | 3.5 years
  Safety will be assessed by Adverse event and Serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: GHIAS UN NABI, FCPS,MRCP, Principal Investigator — PROFESSOR OF MEDICINE
Locations (1):
- Medical Unit 1,Lahore General Hospital,Postgraduate Medical Institute, Lahore, Punjab Province, Pakistan